CLINICAL TRIAL: NCT00757757
Title: A Phase I/II Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MCS110 in Patients With Prostate Cancer and Bone Metastases
Brief Title: A Phase I/II Open-label Study of MCS110 in Patients With Prostate Cancer and Bone Metastases
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMCS110A2101
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer; Bone Metastases
Keywords: Prostate cancer; bone metastases; anti-M-CSF; M-CSF antibody; M-CSF; Prostate Cancer with bone metastases
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MCS110 (Experimental)
  Interventions: Drug: MCS110

INTERVENTIONS:
Drug: MCS110 — Anti-M-CSF antibody

SUMMARY:
This study will evaluate the safety and efficacy of MCS110 in patients with prostate cancer and bone metastases

ELIGIBILITY:
Inclusion Criteria:

* Patients with asymptomatic castrate-resistant prostate cancer with bone metastases who have not received any bisphosphonates in the 12 months prior to enrollment
* 18 years old and over

Exclusion Criteria:

* Plan to be on cytotoxic or biologic therapy during study
* Active dental problems
* Active heart complications
* Active infection
* Patients with moderate to severe swelling due to fluid

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Frequency and characteristics of treatment related dose-limiting-toxicities in dose escalation phase | every cycle - (cycle = 28 days)
Type and frequency of adverse drug reactions and serious adverse drug reactions | every cycle - (cycle = 28 days)

SECONDARY OUTCOMES:
Change in markers of bone resorption and formation (pre- vs. post-treatment) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - NV Cancer Institute, Las Vegas, Nevada
  - CTRC, San Antonio, Texas

REFERENCES:
- See also: Results for CMCS110A2101 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4613